CLINICAL TRIAL: NCT05917769
Title: Comparison of Rocabado Approach Versus Postural Correction Exercises on Kinesiophobia and Interincisal Distance in Patients With Temporo-Mandibular Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/9
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Temporo-mandibular Dysfunction

STUDY DESIGN:
Intervention Model Description: Group A will receive conventional therapy for pain management and Rocabado exercises.
  Group B will receive similar basic conventional therapy for pain management and perform posture correction exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Rocabdo exercises) (Experimental): The exercises created by Dr. Rocabado, will be performed by the patient at home, consist of six different exercises and six repetitions of each exercise, performed six times per day. It consists of Tongue 'Clucking', Controlled TMJ Rotation on Opening, Mandibular Rhythmic Stabilization, Upper Cervical Distraction, Axial Extension of the Cervical Spine and Shoulder Girdle Retraction.
  Interventions: Other: Rocabdo exercises
- Group B (Postural correction exercises) (Experimental): This group will perform posture correction exercises for six days and six times per day. Posture correction exercises include chest stretch , wall stretch , chin tuck in and face down arm lifts.
  Interventions: Other: Postural correction exercises

INTERVENTIONS:
Other: Rocabdo exercises — The exercises created by Dr. Rocabado, will be performed by the patient at home, consist of six different exercises and six repetitions of each exercise, performed six times per day.
  It consists of Tongue 'Clucking', Controlled TMJ Rotation on Opening, Mandibular Rhythmic Stabilization, Upper Cervical Distraction, Axial Extension of the Cervical Spine and Shoulder Girdle Retraction. This group will only perform Rocabdo exercises.
  Arms: Group A (Rocabdo exercises)
Other: Postural correction exercises — * Posture correction exercises will be performed six times a day for six days.
  * Patient will be assessed on the first day and then on the last day of the treatment, i.e., on 6th day the patient will be re-assessed after they have performed posture correction exercises.
  * Posture correction exercises consist of chin tuck in, chest stretch, wall stretch, on your Back chest stretch and face down arm lifts.
  Arms: Group B (Postural correction exercises)

SUMMARY:
Temporo-mandibular dysfunction can cause pain and tenderness of jaw so posture correction exercises and Rocabado exercises will be performed targeting jaw opening and kinesiophobia.

DETAILED DESCRIPTION:
Temporo-mandibular dysfunction refers to pain in area of Temporo-mandibular joint and masticatory muscles.Temporo-mandibular dysfunction can cause pain or tenderness of jaw and aching pain in and around the ear along with difficulty in chewing.In addition to these symptoms the Temporo-mandibular dysfunction results in impairment of mouth opening. So the posture correction exercises and Rocabado exercises will be used to treat patients which will target jaw opening and kinesiophobia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female of 18 to 45 years with TMD pain for less than six months and pain rating at least moderate in severity
* Must not be receiving any treatment for TMD at the onset of the study (for example, an occlusal splint, prescription medication)
* Pain must have been of masticatory muscle origin
* Pain on jaw movement, headache and referred pain are suggestive of a muscular problems.

Exclusion Criteria:

* Patients of Systemic rheumatic disease & Fibromyalgia
* Dental pathology
* Orofacial pain disorders
* Cervical structural pathology
* Current use of analgesics more than 3 days per week
* Current use of narcotics, hypnotic drugs, sedatives, or muscle relaxants

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Mouth opening | 6 days
  Maximum pain free opening from incisor to incisor measured vertically by ruler method where the score of less than 25mm indicate TMJ dysfunction
Kinesiophobia | 6 days
  Kinesiophobia is excessive fear of physical movement that results from a feeling of vulnerability to painful injury Or re-injury where the score of 37 on Tampa scale indicate there is kinesiophobia

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan